CLINICAL TRIAL: NCT06677203
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study of ASN51 in Adults With Early Alzheimer's Disease
Brief Title: Study of ASN51 in Adults With Early Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic decision
Sponsor: Asceneuron S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASN51-201
Record Dates: First submitted 2024-11-05; First posted 2024-11-06 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; ASN51
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- ASN51: Low Dose (Experimental): Participants were to receive low dose of ASN51 orally, once daily (QD) for up to 24 weeks in the double-blind placebo-controlled intervention period or up to 36 weeks long-term extension period.
  Interventions: Drug: ASN51
- ASN51: High Dose (Experimental): Participants were to receive high dose of ASN51 orally, QD for up to 24 weeks in the double-blind placebo-controlled intervention period or up to 36 weeks long-term extension period.
  Interventions: Drug: ASN51
- Placebo (Placebo Comparator): Participants were to receive ASN51 matching placebo orally, QD for up to 24 weeks in the double-blind placebo-controlled intervention period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ASN51 — Oral capsules
  Arms: ASN51: High Dose; ASN51: Low Dose
Drug: Placebo — Oral capsules
  Arms: Placebo

SUMMARY:
The main purpose of this study is to evaluate the safety, tolerability, and effect on biomarkers of disease pathophysiology and pathology, pharmacokinetics (PK), and preliminary effects on measures of clinical efficacy of multiple doses of ASN51 in adult participants with early Alzheimer's disease (AD).

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female age 50 to 80 years.
2. A clinical diagnosis of Alzheimer's disease (AD) at either the mild cognitive impairment or mild AD dementia stage per National Institute on Aging and the Alzheimer's Association, consistent with Stage 3 and Stage 4 in the Food and Drug Administration (FDA) draft guidance for early AD.
3. Mini-Mental State Examination score of 20 to 28 (inclusive).
4. A plasma pTau217 result consistent with the presence of amyloid pathology.
5. Must have a care partner who, in the investigator's judgment, has frequent and sufficient contact with the participant as to be able to provide accurate information about the participant's cognitive and functional abilities. The care partner must be literate and provide informed consent.

Key Exclusion Criteria:

1. Any medical or neurological/neurodegenerative condition (other than AD) that, in the opinion of the Investigator, might be a contributing cause to the participant's cognitive impairment (e.g., current history of substance abuse, uncontrolled vitamin B12 deficiency or abnormal thyroid function, stroke or other cerebrovascular condition, normal pressure hydrocephalus, Parkinson's Disease, Lewy body dementia, cerebral amyloid angiopathy, frontotemporal dementia) or could lead to discontinuation, lack of compliance, interference with study assessments, or safety concerns.
2. Non-amnestic presentation of AD as judged by the investigator.
3. Woman of childbearing potential.
4. Any prior or ongoing exposure to active or passive anti-amyloid immunotherapy, anti-tau immunotherapy, an anti-tau antisense oligonucleotide or gene therapy, or O-linked-β-N-acetylglucosaminidase (O-GlcNAcase) inhibitor.

Other protocol defined inclusion and exclusion criteria could apply.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-11-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - K2 Medical Research, Clermont, Florida
  - K2 Medical Research - The Villages, Lady Lake, Florida
  - K2 Medical Research, Maitland, Florida
  - Alzheimer's Treatment and Research Center, Stuart, Florida
  - Alzheimer's Treatment and Research Center, Wellington, Florida
  - Columbus Memory Center, LLC, Columbus, Georgia
  - Re:Cognition Health, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 123 participants with Alzheimer's disease (AD) were enrolled in the study. The study was terminated due to a strategic decision by the sponsor before randomization and hence no participants received treatment, and no data were collected or evaluated for this study.
Groups:
- ASN51 Low Dose: Participants were to receive low dose of ASN51 orally, once daily (QD) for up to 24 weeks in the double-blind placebo-controlled intervention period or up to 36 weeks long-term extension period.
- ASN51 High Dose: Participants were to receive high dose of ASN51 orally, QD for up to 24 weeks in the double-blind placebo-controlled intervention period or up to 36 weeks long-term extension period.
Period: Overall Study
Arm/Group | ASN51 Low Dose | ASN51 High Dose | Placebo
Started | 0 | 0 | 0
Completed | 0 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The study was terminated due to a strategic decision by the sponsor. No participants received treatment, and no data were collected or evaluated for this study.
Groups:
- ASN51 Low Dose: Participants receive low dose of ASN51 orally, QD for up to 24 weeks in the double-blind placebo-controlled intervention period or up to 36 weeks long-term extension period.
- Total: Total of all reporting groups
Arm/Group | ASN51 Low Dose | ASN51 High Dose | Placebo | Total
Number analyzed (Participants) | 0 | 0 | 0 | 0
Age, Continuous
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)
Region of Enrollment [unit: participants]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related.
Time Frame: From first dose up to end of the study up to Week 28
Population: as for baseline characteristics
Groups:
- ASN51 Low Dose: Participants were to receive low dose of ASN51 orally, QD for up to 24 weeks in the double-blind placebo-controlled intervention period or up to 36 weeks long-term extension period.
Arm/Group | ASN51 Low Dose | ASN51 High Dose | Placebo
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Change From Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: C-SSRS is used to assess the suicidality of participants and assessment includes "yes" or "no" responses for 5 questions, each related to suicidal ideation and suicidal behavior. Numeric ratings are provided for suicidal ideation (score ranges from 1 to 5, where higher scores indicate more suicidal ideation) and suicidal behavior (score ranges from 0 to 4 where higher total scores indicate more suicidal behavior).
Time Frame: Baseline up to Week 28
Population: as for baseline characteristics
Arm/Group | ASN51 Low Dose | ASN51 High Dose | Placebo
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Change From Baseline in Cerebrospinal Fluid (CSF) Plasma Tau Phosphorylated at Threonine-217 (pTau217) Through Week 24
Time Frame: Baseline through Week 24
Population: as for baseline characteristics
Arm/Group | ASN51 Low Dose | ASN51 High Dose | Placebo
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in CSF Total Tau Protein Through Week 24
Time Frame: Baseline through Week 24
Population: as for baseline characteristics
Arm/Group | ASN51 Low Dose | ASN51 High Dose | Placebo
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Change From Baseline in Plasma pTau217 Through Week 24
Time Frame: Baseline through Week 24
Population: as for baseline characteristics
Arm/Group | ASN51 Low Dose | ASN51 High Dose | Placebo
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Change From Baseline in MK-6240 Tau Positron Emission Tomography (PET) Signal Through Week 24
Time Frame: Baseline through Week 24
Population: as for baseline characteristics
Arm/Group | ASN51 Low Dose | ASN51 High Dose | Placebo
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Trough Plasma Concentration (Cmin) of ASN51 in Plasma at Steady State
Time Frame: Pre-dose on Day 1 and at multiple time points post-dose up to Week 24
Population: as for baseline characteristics
Arm/Group | ASN51 Low Dose | ASN51 High Dose | Placebo
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Maximum Plasma Concentration (Cmax) of ASN51 at Steady State
Time Frame: Pre-dose on Day 1 and at multiple time points post-dose up to Week 24
Population: as for baseline characteristics
Arm/Group | ASN51 Low Dose | ASN51 High Dose | Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs were not collected in this study.
Description: The study was terminated due to a strategic decision by the sponsor. No participants received treatment, and no data were collected or evaluated for this study.
Groups:
- ASN51 10 mg: Participants received 10 mg of ASN51 orally, QD for up to 24 weeks in the double-blind placebo-controlled intervention period or up to 36 weeks long-term extension period.
- ASN51 20 mg: Participants received 20 mg of ASN51 orally, QD for up to 24 weeks in the double-blind placebo-controlled intervention period or up to 36 weeks long-term extension period.
- Placebo: Participants received ASN51 matching placebo orally, QD for up to 24 weeks in the double-blind placebo-Controlled intervention period.
Arm/Group | ASN51 10 mg | ASN51 20 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
The study was terminated due to a strategic decision by the sponsor. No participants received treatment, and no data were collected or evaluated for this study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement finally allows PI to publish independently.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-10-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT06677203/Prot_SAP_000.pdf